CLINICAL TRIAL: NCT00304226
Title: A 14 Week Study to Evaluate Effectiveness of a Valsartan Versus an Amlodipine Treatment Strategy in Achieving Blood Pressure Control in Patients With Stage 1 or Stage 2 Hypertension or Uncontrolled on Present Monotherapy
Brief Title: Effectiveness of a Valsartan Based Versus an Amlodipine Based Treatment Strategy in naïve Patients With Stage 1 or Stage 2 Hypertension or in Patients Uncontrolled on Current Monotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAH631B2406
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension
Keywords: Valsartan,; amlodipine,; hydrochlorothiazide
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Amlodipine

INTERVENTIONS:
Drug: valsartan
Drug: amlodipine

SUMMARY:
The population for this current study will include stage 1 and stage 2 hypertensive patients who are newly diagnosed or didn't have treatment during the last 3 months and patients who are currently treated but uncontrolled on present monotherapy.

The purpose of this study is to evaluate the efficacy of a treatment with valsartan versus a treatment with amlodipine in reaching blood pressure control after 14 weeks of treatment.

ELIGIBILITY:
Inclusion criteria Stage/grade 1 or stage/ grade 2 hypertension, MSSBP ≥ 140 mm Hg, and/ or MSDBP ≥ 90 mm Hg, at Visit 1 and 2 in untreated patients Or Patients who are currently treated on monotherapy and uncontrolled and have a blood pressure ≤ 160/100 mm Hg at Visit 1 and Visit 2

Exclusion criteria Current treatment with a CCB MSSBP ≥ 180 mm Hg or MSDBP ≥ 110 mm Hg at any time between visit 1 and Visit 2 History of hypersensitivity to any of the study drugs or to drugs with similar chemical structures Evidence of a secondary form of hypertension Cerebrovascular accident or myocardial infarction during the last 12 months, prior to Visit 1 Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1288 (Actual)
Dates: Start 2006-02; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure less than 140/90 mmHg after 14 weeks

SECONDARY OUTCOMES:
Blood pressure less than 140/90 mmHg after 4, 8, and 11 weeks
Blood pressure less than 140/90 mmHg after 4, 8, 11, and 14 weeks
Time when blood pressure reaches less than 140/90 mmHg
Change in blood pressure at baseline, week 4, 8, 11, and 14
Adverse events and serious adverse events at each study visit for 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novatis Pharmaceuticals
Locations (2):
- Investigative Centers, Germany
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Result] Zappe D, Papst CC, Ferber P; PROMPT Investigators. Randomized study to compare valsartan +/- HCTZ versus amlodipine +/- HCTZ strategies to maximize blood pressure control. Vasc Health Risk Manag. 2009;5:883-92. doi: 10.2147/vhrm.s8062. Epub 2009 Nov 2. PMID 19898644